CLINICAL TRIAL: NCT03807505
Title: Erector Spinae Plane Versus Interscalene Blocks for Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 48351
Record Dates: First submitted 2018-12-14; First posted 2019-01-17 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Anesthesia, Local; Phrenic Nerve Paralysis; Upper Extremity Injury; Shoulder Injury
MeSH Terms: conditions — Arm Injuries; Shoulder Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interscalene nerve block (Active Comparator): Patients undergoing rotator cuff repair surgery or total shoulder arthroplasty will undergo a single shot interscalene brachial plexus nerve block or an interscalene brachial plexus nerve catheter. In the preoperative area, all participants will be asked baseline indicators of pain level via a Numeric Rating Scale (NRS, 0-10, where 0 is no pain and 10 is the worst imaginable pain) and diaphragmatic excursion will be measured bilaterally using ultrasonography before nerve block placement. Motor and sensory exams will also be performed. The same parameters will be measured 30 minutes after the block is performed. In the recovery room, those with nerve catheters will receive a dose of local anesthetic. All patients will have the same parameters measured 30 minutes postoperatively.
  Interventions: Procedure: Interscalene brachial plexus nerve block
- Erector Spinae Plane block (Active Comparator): Patients undergoing rotator cuff repair surgery or total shoulder arthroplasty will undergo a single shot erector spinae plane block or receive erector spinae plane catheter. In the preoperative area, all participants will be asked baseline indicators of pain level via a Numeric Rating Scale (NRS, 0-10, where 0 is no pain and 10 is the worst imaginable pain) and diaphragmatic excursion will be measured bilaterally using ultrasonography before nerve block placement. Motor and sensory exams will also be performed. The same parameters will be measured 30 minutes after the block is performed. In the recovery room, those with nerve catheters will receive a dose of local anesthetic. All patients will have the same parameters measured 30 minutes postoperatively.
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Interscalene brachial plexus nerve block — An interscalene brachial plexus nerve block (single shot or catheter, depending on surgical procedure) will be placed under ultrasound guidance and all patients will receive 10cc 0.5% ropivacaine during block placement. Patients with a nerve catheter will receive a bolus of 5cc 0.5% ropivicaine postoperatively, on arrival to the recovery unit.
  Arms: Interscalene nerve block
Procedure: Erector spinae plane block — An erector spinae plane block (single shot or catheter, depending on surgical procedure) will be placed under ultrasound guidance and all patients will receive 10cc 0.5% ropivacaine during block placement. Patients with a nerve catheter will receive a bolus of 5cc 0.5% ropivicaine postoperatively, on arrival to the recovery unit.
  Arms: Erector Spinae Plane block

SUMMARY:
The goal of this study is the evaluation of erector spinae plane (ESP) blocks as an alternative to interscalene brachial plexus nerve blocks for rotator cuff repair and total shoulder arthroplasty procedures. Currently, single shot interscalene nerve blocks are performed for rotator cuff repair surgeries, and interscalene nerve catheters are placed for total shoulder arthroplasty surgeries. Erector spinae plane blocks are commonly used as part of the anesthetic plan for other surgeries, but less so for shoulder surgeries. The investigators would like to study whether an ESP block can provide similar pain control compared to an interscalene nerve block, with less risk of upper extremity motor block and phrenic nerve block.

ELIGIBILITY:
Inclusion Criteria:

- All adult patients (18 years and over) scheduled for rotator cuff surgery or total shoulder arthroplasty surgery requiring a nerve block as part of their anesthetic care

Exclusion Criteria:

* concomitant life-threatening injuries and other concomitant injuries causing significant pain.
* pregnancy,
* any condition impairing patient's ability to consent to participation in study
* an existing condition contraindicating a nerve block, i.e. nerve injury, existing bleeding disorder
* infection in the vicinity of the block, and patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of diaphragmatic paresis or paralysis | Before block placement, and 30 minutes after catheter is bolused in recovery
  Change in diaphragmatic excursion (measured bilaterally using ultrasonography) from before block placement to 30 minutes after catheter is bolused in recovery
Pain score | 48 hours
  Pain scores for all patients will be recorded through the first 48 hours postoperatively using the Numeric Rating scale (ranging from 0 to 10, 0 is no pain and 10 is the worst imaginable pain).

SECONDARY OUTCOMES:
Brachial plexus sensory exam change | Before block placement, and 30 minutes after catheter is bolused in recovery
  Brachial plexus sensory exam change: dichotomous measurement (yes or no) for change in sensation over C5-C8 dermatomes
Brachial plexus motor exam change | Before block placement, and 30 minutes after catheter is bolused in recovery
  Brachial plexus motor exam change: dichotomous measurement (yes or no) for change in finger extension, finger abduction and thumb opposition to resistance
Opioid Consumption | 48 hours
  Opioid consumption in the recovery room and in the first 48 hours postoperatively will be recorded
Adverse effects | 72 hours
  Patient-reported adverse effects (dichotomous measure, yes/no): dyspnea, Horner syndrome, hoarseness, difficulty participating in physical therapy due to block
Patient satisfaction | 72 hours
  Patient satisfaction with the nerve block (dichotomous measure: yes/no)
Incentive spirometry volume change | 24 hours
  Change in incentive spirometry volume from baseline (prior to block) to recovery room, and to postoperative day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Ban Tsui, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care (SHC), Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Urmey WF, Talts KH, Sharrock NE. One hundred percent incidence of hemidiaphragmatic paresis associated with interscalene brachial plexus anesthesia as diagnosed by ultrasonography. Anesth Analg. 1991 Apr;72(4):498-503. doi: 10.1213/00000539-199104000-00014. PMID 2006740
- [Background] Riazi S, Carmichael N, Awad I, Holtby RM, McCartney CJ. Effect of local anaesthetic volume (20 vs 5 ml) on the efficacy and respiratory consequences of ultrasound-guided interscalene brachial plexus block. Br J Anaesth. 2008 Oct;101(4):549-56. doi: 10.1093/bja/aen229. Epub 2008 Aug 4. PMID 18682410
- [Background] Tsui BCH, Fonseca A, Munshey F, McFadyen G, Caruso TJ. The erector spinae plane (ESP) block: A pooled review of 242 cases. J Clin Anesth. 2019 Mar;53:29-34. doi: 10.1016/j.jclinane.2018.09.036. Epub 2018 Oct 3. PMID 30292068
- [Background] Tsui BCH, Mohler D, Caruso TJ, Horn JL. Cervical erector spinae plane block catheter using a thoracic approach: an alternative to brachial plexus blockade for forequarter amputation. Can J Anaesth. 2019 Jan;66(1):119-120. doi: 10.1007/s12630-018-1170-7. Epub 2018 Jun 4. No abstract available. PMID 29868941
- [Background] Forero M, Rajarathinam M, Adhikary SD, Chin KJ. Erector spinae plane block for the management of chronic shoulder pain: a case report. Can J Anaesth. 2018 Mar;65(3):288-293. doi: 10.1007/s12630-017-1010-1. Epub 2017 Nov 13. PMID 29134518
- [Derived] Sun LY, Basireddy S, Gerber LN, Lamano J, Costouros J, Cheung E, Boublik J, Horn JL, Tsui BCH. Continuous interscalene versus phrenic nerve-sparing high-thoracic erector spinae plane block for total shoulder arthroplasty: a randomized controlled trial. Can J Anaesth. 2022 May;69(5):614-623. doi: 10.1007/s12630-022-02216-1. Epub 2022 Mar 2. PMID 35237953